CLINICAL TRIAL: NCT01181518
Title: Observational Study: Biomarker Research for Tamoxifen Pharmacogenetics Among Asian Breast Cancer Patients
Brief Title: Tamoxifen Pharmacogenetics in Asian Breast Cancer Women
Acronym: Tamoxifen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Professor, Inje University
Other Study IDs: 09-140
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Poisoning by, Adverse Effect of and Underdosing of Tamoxifen
Keywords: Tamoxifen; Pharmacogenomics; Breast cancer
MeSH Terms: conditions — Poisoning; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples for genotyping and pharmacokinetic analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinical outcome of tamoxifen treatment in breast cancer patients may be influenced by the activity of cytochrome P450 enzymes involving in tamoxifen biotransformation.

DETAILED DESCRIPTION:
The investigators investigated the prognostic and/or predictive value of genetic polymorphisms of enzymes involved in tamoxifen metabolism for the treatment outcome among Asian breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* incident breast cancer patients who underwent surgery

Exclusion Criteria:

* previous cancer history before breast cancer diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who underwent surgery at Busan Paik Hospital, Inje University
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Association between genetic polymorphisms of CYP2D6, CYP2C19, and CYP3A5 and disease free survival among tamoxifen treated breast cancer patients | five years
  Association between genetic polymorphisms of CYP2D6, CYP2C19, and CYP3A5 and disease free survival among tamoxifen treated breast cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: JaeGook Shin, MD,PhD, Principal Investigator — Inje University
Locations (1):
- Inje University, Busan, Busan, South Korea